CLINICAL TRIAL: NCT04527068
Title: QL1101A,a Biosimilar of Bevacizumab,in Combination With JS001,a Anti-pd-1 Antibody in Patients With pMMR/MSS Refractory Metastatic Colorectal Cancer: a Single-arm,Open-Label, Prospective, Single-center Study
Brief Title: QL1101 in Combination With JS001 in Patients With pMMR/MSS Refractory Metastatic Colorectal Cancer
Acronym: BEVTOR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry); Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEVTOR202008
Record Dates: First submitted 2020-08-23; First posted 2020-08-26 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-08

CONDITIONS: Refractory Metastatic Colorectal Cancer; pMMR; MSS
Keywords: metastatic colorectal cancer; refractory; QL1101; JS001; tripleitriumab; bevacizumab; pMMR; MSS; immunotherapy; PD-1; VEGF; antiangiogenic; mCRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bevacizumab +Tripleitriumab (Experimental): Participants receive bevacizumab 7.5mg/kg and tripleitriumab 240mg in day 1 intravenously every 3week until disease progression or unacceptable toxicity
  Interventions: Drug: Bevacizumab; Drug: Tripleitriumab

INTERVENTIONS:
Drug: Bevacizumab — 7.5 mg/kg intravenously every 3week
  Other Names: QL1101
Drug: Tripleitriumab — 240mg intravenously every 3week
  Other Names: JS001

SUMMARY:
This is a single-arm,open-label, prospective, single-center Study of QL1101 and JS001 in patients with pMMR/MSS refractory metastatic colorectal cancer.

QL1101 is a biosimilar of bevacizumab (Avastin) produced and provided by Qilu Pharmaceutical Co., Ltd., which has been marketed in China.It's a humanized monoclonal IgG1 antibody prepared by recombinant DNA technology. By binding to human vascular endothelial growth factor (VEGF), it inhibits the binding of VEGF to its receptor, blocks the signal transduction pathway of angiogenesis, and inhibits tumor cell growth. Be produced and provided by Shanghai Junshi Bioscience Co., Ltd. ,JS001(Tripleitriumab) is the first China-developed humanized monoclonal antibody against programmed death 1 (PD-1) approved for marketing in China.

Antiangiogenic drugs combined with PD-1 monoclonal antibodies may reverse the insensitivity of pMMR/MSS refractory colorectal cancer to PD-1 inhibitors.

The primary objective of this study is to investigate the safety and efficacy of the subjects who given the combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unresectable advanced (metastatic or locally advanced) colorectal cancer confirmed by histology or cytology
2. The results of tissue samples or liquid biopsy measured by the pathology department or laboratory department of a tertiary hospital and a qualified genetic testing company meet any of the following:

   1. The test result of immunohistochemistry is mismatch repair protein integrity (pMMR)
   2. The test result of NGS or liquid biopsy + NGS is MSI-L or MSS
   3. The test result of PCR is MSI-L or MSS
3. Previous treatment must meet all of the following conditions:

   1. Thymidylate synthase inhibitors,such as 5-FU, capecitabine, UFT,raltitrexed,Tegafur,Gimeracil and Oteracil Porassium Capsules,have been accepted for disease metastasis or as adjuvant therapy. Thymidylate synthase inhibitors can be combined with oxaliplatin or irinotecan
   2. Have received the irinotecan-containing regimen (single or combination) for the treatment of metastatic tumors and the treatment has failed, or has a record of unsuitable irinotecan-containing regimen treatment

      * Failure is defined as disease progression (clinical or radiological) or intolerance to irinotecan-containing regimens. Intolerance is defined as discontinuation of use due to any of the following reasons: severe allergic reaction or delayed recovery from toxicity, which prevents retreatment
      * Recorded conditions that are not suitable for irinotecan treatment include (but are not limited to) known hypersensitivity to irinotecan, abnormal glucuronidation of bilirubin, Gilbert syndrome, or received pelvic or abdominal radiation therapy.
   3. Has received the oxaliplatin-containing regimen (single or combination) for the treatment of metastatic tumors and the treatment has failed, or recurred within 6 months after completion of oxaliplatin-containing adjuvant therapy,or has a record of unsuitable oxaliplatin-containing regimen treatment

      * Failure is defined as disease progression (clinical or radiological) or intolerance to oxaliplatin-containing regimens, where intolerance is defined as discontinuation of use due to any of the following reasons: severe allergic reaction, persistent severe neurotoxicity or delayed recovery of toxicity prevents retreatmen
      * Recorded conditions that are not suitable for treatment with oxaliplatin-containing regimens include but are not limited to known hypersensitivity to oxaliplatin or other platinum compounds, renal insufficiency, or sensory neuropathy of grade ≥2
   4. For patients with RAS wild type colorectal cancer: patients who have received cetuximab or panizumab regimens (monotherapy or combination) for tumor metastasis and failed, or have been recorded to be unsuitable for treatment with cetuximab or panizumab regimens

      * Failure is defined as disease progression (clinical or radiological) or intolerance to cetuximab or panizumab therapy, where intolerance is defined as discontinuation of use due to any of the following reasons: severe infusion reaction, delayed recovery of persistent skin toxicity or toxicity, preventing retreatment
      * Recorded conditions that are not suitable for treatment with regimens containing cetuximab or panitumumab include (but are not limited to) allergy to cetuximab or activated RAS or RAF mutations
   5. Patients are allowed to receive previous VEGF targeted therapy, such as bevacizumab, aflibercept, ramolumab, rigofenib or fuquitinib, and to receive immune checkpoint inhibitors such as PD-1 / PD-L1 antibodies or CTLA-4 antibodies other than tripleitriumab, but not to receive anti-angiogenic drugs in combination with immune checkpoint inhibitors
   6. Allow patients to be previously treated with TAS-102
4. Age ≥18 and ≤75 years old
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 ~ 2
6. At least one measurable lesion have been the confirmatory detection respect to RECIST version 1.1
7. Life expectancy ≥ 3 months
8. Subjects must have normal organ and marrow function as defined belowno blood transfusion and blood products within 2 weeks before screening, no use of hematopoietic stimulating factors, and test results within 7 days before the registration date are recognized):

   1. Blood routine examination standards：

      * WBC≥3.0 × 10^9/L
      * Hb ≥80 g/L
      * ANC ≥ 1.5×10^9/L
      * PLT ≥ 100×10^9/L
   2. Liver function test standards:

      * TBIL≤1.5 times the upper limit of normal（ULN）, the TBIL of patients with Gilbert's syndrome < 4×ULN
      * ALT and AST ≤2.5×ULN，If liver metastasis is present，ALT and AST≤5×ULN
   3. Kidney function test standards:

      * SCr≤1.5×ULN，or Creatinine clearance >50ml/min（Creatinine clearance can be directly measured by 24-hour urine sampling or calculated by the following Cockcroft-Gault formula:Female GFR =1.04×(140-age）× weight(kg)/SCr（μmol/L）,Male GFR=1.23×(140-age）× weight(kg)/SCr（μmol/L）
      * The results of routine urine test showed that urinary protein <2 +. When the urine routine test shows that the urine protein is ≥ 2 + at baseline, 24-hour urine should be collected and the result of protein content < 1g
   4. Coagulation function: Within 7 days before treatment, the international standardized ratio (INR) ≤ 1.5 (if anticoagulants are used, INR ≤ 3.0), prothrombin time ((PT)) and activated partial thromboplastin time ((APTT)) ≤ 1.5 × ULN
   5. Color Doppler echocardiography: Left ventricular ejection fraction ((LVEF)) ≥ 55%
   6. 12-lead ECG: QT interval (QTcF) < 470 msec corrected by Fridericia method
9. Subjects can understand and voluntarily participate in this study, sign informed consent, have good compliance, and cooperate with follow-up
10. Female subjects of childbearing age, male subjects and partners of male subjects agreed to use reliable contraceptive methods (such as abstinence, sterilization, contraceptive, contraceptive medroxyprogesterone injection or subcutaneous implantation of contraception, etc.) during the study period and within 6 months after experimental drug infusion.

Exclusion Criteria:

1. Have received any systemic chemotherapy within 28 days before the first study drug, or have received immunotherapy (such as interleukin, interferon, thymosin), hormone therapy, targeted therapy, or any research therapy within 14 days or 5 half-lives before the first study drug, whichever is the shorter, but immune checkpoint inhibitors are allowed to be pretreated
2. Received any Chinese herbal medicine or proprietary Chinese medicine for cancer control within 14 days prior to the use of the drug for the first study
3. Patients with primary malignancies other than bowel cancer within 5 years before randomization, except for fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical resection,ductal carcinoma in situ after radical resection,and papillary thyroid cancer
4. Patients whose toxicity and side effects (due to previous anticancer treatments) have not returned to baseline or stable levels, unless such AE is not considered to pose safety risks (such as hair loss, neuropathy and abnormal results of specific laboratory tests)
5. Uncontrolled hypertension after treatment (systolic blood pressure ≥ 140mmHg and / or diastolic blood pressure ≥ 90mmHg). Have a history of hypertensive crisis or hypertensive encephalopathy
6. Any unstable systemic diseases: including but not limited to cerebrovascular accidents (transient ischemic attack, cerebral hemorrhage, cerebral infarction, etc. within 6 months before screening), deep vein thrombosis, cardiogenic chest pain (moderate pain in the 28 days before screening leads to instrumental limitation of activities of daily living), myocardial infarction (within 6 months before screening), coronary angioplasty or history of stent placement (within 6 months before screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ grade III within 6 months before screening), symptomatic pulmonary embolism (within 28 days before screening) ), ventricular arrhythmia events with severity ≥ 2 (within 6 months before screening), syncope, seizures or falls (within 28 days before screening), poorly controlled diabetes or poorly controlled electrolyte disorders
7. Clinically significant third space effusion (such as a large amount of pleural effusion, ascites, pericardial effusion that cannot be controlled by pumping or other treatments)
8. Symptomatic central nervous system metastasis; patients with asymptomatic brain metastasis or stable symptoms after brain metastasis can participate in this study as long as they meet all the following criteria: there are measurable lesions outside the central nervous system; no midbrain, pons, cerebellum, medulla oblongata or spinal cord metastasis; no previous history of intracranial hemorrhage
9. The following medical history within 6 months before screening: peptic ulcer, gastrointestinal perforation, corrosive esophagitis or gastritis, inflammatory bowel disease or diverticulitis, abdominal fistula, or intra-abdominal abscess
10. Patients with tracheo-esophageal fistula
11. Patients with partial or complete bowel obstruction
12. Untreated patients with chronic hepatitis B or chronic hepatitis B virus (HBV) carriers with HBV DNA > 500IU/mL (or the lower limit of detection) and patients with hepatitis C virus (HCV) RNA positive should be excluded. Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B (HBVDNA <500IU/mL or the lower limit of detection) and cured hepatitis C patients can be selected
13. Human immunodeficiency virus (HIV) antibodies or syphilis testing positive
14. Severe chronic or active infections (according to CTCAE version 5.0, ≥ grade 3) require systemic antibacterial, antifungal or antiviral treatment, including tuberculosis j infections. Patients with a history of active tuberculosis infection ≥ 1 year before screening should also be excluded, unless proof can be provided that appropriate treatment has been completed
15. Patients with Child - Pugh B or more severe liver cirrhosis
16. Severe unhealed wound ulcers or fractures, or major surgery within 6 weeks before enrollment or expected major surgery during the study period; minor surgery within 48 hours before receiving the study drug for the first time (outpatient or inpatient surgery requiring local anesthesia，including central venipuncture catheterization); the current or recent (within 10 days before the first dose of study medication) use of aspirin for 10 days (> 325 mg/day) or other known to inhibit platelet function of NASIDS;the current or recent (within 10 days before receiving the first study drug) use of full-dose oral or parenteral anticoagulants or thrombolytic agents, but prophylactic use of anticoagulants is allowed; have hereditary bleeding tendencies or coagulation disorders (e.g. hemophilia, coagulopathy, thrombocytopenia, etc.), or a history of thrombosis
17. Currently suffering from interstitial lung disease or CT showing active pneumonia during screening
18. History of active autoimmune disease or autoimmune disease that may recur

    NOTE: Patients with the following diseases will not be excluded for the time being, and further screening may be carried out:
    1. Well-controlled type I diabetes
    2. HypothyroidismHypothyroidism (only hormone replacement therapy is needed for treatment)
    3. Well-controlled celiac disease
    4. Skin diseases that do not require systemic treatment (eg vitiligo, psoriasis, hair loss)
    5. Any other diseases that are not expected to recur without external triggers
19. Patients with a history of allergic disease or allergic constitution
20. Suffer from any disease that requires corticosteroids (dose of prednisone or equivalent drugs> 10 mg/day) or other immunosuppressive drugs for systemic treatment within ≤ 14 days before the first study drug administration

    NOTE: patients who have used any of the following steroid treatments do not need to be excluded:
    1. Steroids are used to replace adrenal function (prednisone or equivalent dose ≤ 10mg/ day)
    2. Local, ocular, intra-articular, intranasal or inhaled corticosteroids with very low systemic absorption
    3. Short-term (≤ 7 days) prophylactic use of corticosteroids (e.g. for contrast medium allergy) or for the treatment of non-autoimmune diseases (e.g. delayed type hypersensitivity caused by contact allergens)
21. History of primary immunodeficiency, or history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation, or history of grade 3 to 4 immune-mediated toxicity caused by other immunotherapy
22. Patients with a history of allergy to studied drugs or similar drugs or excipients
23. Patients with a history of alcohol or drug abuse who cannot be cured or who have mental disorders
24. Vaccination with live attenuated vaccine within 28 days before screening (including but not limited to measles, mumps and rubella vaccines, live attenuated influenza vaccine (nasal), varicella vaccine, oral polio vaccine, rotavirus vaccine, yellow fever vaccine,BCG, typhoid vaccine and typhus vaccine)
25. Pregnant or lactating women or women preparing to become pregnant or breastfeeding during the study
26. Other conditions that researchers consider inappropriate for inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-20 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From the first use of research drugs to documented disease progression per RECIST 1.1 and iRECIST or death from any cause, whichever occurs first, assessed up to 18 months
  Will be estimated using the Kaplan-Meier method, and Cox proportional hazards models will be used to estimate the treatment hazard ratios. PFS will use a logrank test stratified on the randomization stratification factors with a one-sided type I error rate of 2.5%.

SECONDARY OUTCOMES:
Overall survival (OS) | From the first use of research drugs to death from any cause, assessed up to 18 months
  Will be estimated using the Kaplan-Meier method, and Cox proportional hazards models will be used to estimate the treatment hazard ratios. OS will be tested at the one-sided 10% level.
Overall response rate(ORR) | up to 18 months
  Best objective response will be evaluated via RECIST 1.1 and iRECIST criteria. Will be compared using Fisher's exact tests with a one-sided type I error rate of 2.5%; multivariable logistic regression modeling will be used to adjust for the effect of any covariates that are associated with these categorical outcomes.
Disease Control Rate (DCR) | up to 18 months
  Disease control is defined as maintaining Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) as the tumor assessment result during the defined time window. DCR (percentage) is defined as number of patients with success of disease control divided by total number of patients in the analysis population multiplied by 100, excluding patients who refuse treatment before the initiation of any treatment. CR: Disappearance of all evidence of disease, PR: Regression of measurable disease and no new sites, PD: Any new lesion or increase by ≥50% of previously involved sites from nadir, SD: Neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for PD taking as reference the MSD
Duration of Response (DOR) | From the date of first tumor assessment with the response status being CR or PR to the date of 1st documented progressive disease, assessed up to 12 months
  The distribution of DOR by treatment group will be estimated using the method of Kaplan-Meier. Six and 12 month durable response (i.e. maintaining CR or PR without progressive disease [PD]) rates by treatment group with confidence intervals will be estimated based on Kaplan-Meier curves. The HR with confidence interval will be estimated based on stratified Cox models (stratified by levels of stratification factors), without and with adjusting for baseline clinical/pathological factors.CR: Disappearance of all evidence of disease, PR: Regression of measurable disease and no new sites, PD: Any new lesion or increase by ≥50% of previously involved sites from nadir

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, M.D., Principal Investigator — The Second Affiliated Hospital of Medical College of Zhejiang University
Locations (1):
- the Second Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No